CLINICAL TRIAL: NCT00964600
Title: Evaluation of the Effect of Bilateral Transversus Abdominis Plane Block on Postoperative Pain Intensity and Analgesia Consumption After Elective Cesarean Delivery
Brief Title: Bilateral Transversus Abdominis Plane Block and Postoperative Pain Intensity After Elective Cesarean Delivery
Acronym: TAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Laleh Eslamian, MD ,associate Prof
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 825
Record Dates: First submitted 2009-08-20; First posted 2009-08-25 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Postoperative Pain
Keywords: transversus abdominis block; postoperative pain; cesarean
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP blockade (Experimental): bilateral TAP blockade at the end of cesarean delivery
  Interventions: Procedure: TAP blockade
- No TAP (No Intervention): These patients would have usual analgesic drugs after cesarean

INTERVENTIONS:
Procedure: TAP blockade — 15 cc Bupivacaine 0.25% ,injected bilaterally in the TAP blockade arm
  Arms: TAP blockade

SUMMARY:
The patients planned to go under elective cesarean delivery under general anesthesia are randomly assigned to have either bilateral transversus abdominis plane (TAP) block or usual standard analgesics after cesarean. Pain score (Verbal Analog Scale VAS) and analgesic requirements are recorded. It's supposed that both are significantly reduced in patients undergoing TAP block.

ELIGIBILITY:
Inclusion Criteria:

1. Elective cesarean delivery
2. Term pregnancies
3. General anesthesia
4. Pfannenstiel incision

Exclusion Criteria:

1. No history of sensitivity to prescribed analgesic (Bupivacaine or related substances)
2. No preeclampsia
3. No history of psychologic disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity after cesarean section | one year

SECONDARY OUTCOMES:
Analgesic prescribed measurement | one year

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Eslamian, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Sharati hospital, Tehran, Tehran Province, Iran